CLINICAL TRIAL: NCT07239089
Title: Outcomes of Endovascular Atherectomy in Femoropopliteal Arterial Disease
Brief Title: Oucomes of Endovascular Atherectomy in Femoropopliteal Arterial Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Ahmed Mohamed Elshimy, Outcomes of Endovascular Atherectomy in femoropopliteal arterial disease, Assiut University
Other Study IDs: AssiutU
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Threatening Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- sample size is 60 patients (30 in each group).
  Interventions: Device: Endovascular Atherectomy

INTERVENTIONS:
Device: Endovascular Atherectomy — Endovascular Atherectomy in femoropopliteal arterial disease

SUMMARY:
Peripheral artery disease (PAD) affects >200 millionadults worldwide and is amajor cause of morbidity ranging from exertional lower extremity pain to ischemic rest pain and ulcer formation.

Endovascular treatment options for PAD have increased dramatically in the past several decades. The traditional endovascular treatment of severe PAD has been balloon angioplasty with or without adjunctive stenting.

The outcomes of balloon angioplasty and stenting are acceptable for short lesion lengths in the superficial femoral artery (SFA) and proximal popliteal arteries.Therefore, there is an established need for technologies that can adequately treat more complex femoropopliteal lesions.

Endovascular atherectomy has emerged as a novel technique for atheroma removal in patients with disease of the SFA or popliteal arteries. Atherectomy offers the advantages of surgical endarterectomy by removing atherosclerotic plaque while remaining a minimally invasive and percutaneous treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients present with CLTI due to femoropopliteal artery disease with the following criteria:

  * Denovo or Recoil
  * Stenosis or occlusion

Exclusion Criteria:

* Patients present with:

  * Previous ipsilateral bypass surgery
  * In-stent restenosis or previous atherectomy
  * Known hypercoagulable disorder or non-atherosclerotic vasculopathy
  * Severe renal insufficiency (eGFR <30) not on dialysis
  * Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the estimated minimum required sample size is 60 patients (30 in each group).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2027-10-22 (Estimated)

PRIMARY OUTCOMES:
Technical success | From october 2025 to october 2027
  completion of the endovascular procedure without the need for further intervention for revascularization and an absence of substantial or complete occlusion in SFA at final angiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Ţahţā, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided